CLINICAL TRIAL: NCT04745858
Title: Compare Bowen's Technique and Muscle Energy Technique on Hamstrings Tightness in Chronic Non-Specific Low Back Pain Patients
Brief Title: Bowen's Technique and Muscle Energy Technique on Hamstrings Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00867 Ateeqa Younis
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: physical therapy; Hamstring; flexibility; Muscle Energy Technique
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen's Technique (Experimental): Sequence of short gentle moves are applied over Hamstrings.Skin slack is taken to lateral side of muscle. The muscle is hooked by the thumbs from its lateral edge. Skin is carried along and thumb is flattened in a medial direction, the muscle plucks under the thumbs. Three alternate sessions per week are be given for 4 weeks. The treatment time for each session is 20 minutes.
  Interventions: Other: Bowen's Technique
- Muscle Energy Technique (Active Comparator): Isometric contraction of hamstrings is performed by the patient being employing 20% of the strength. This contraction is resisted by the practitioner for 7-10 s. A three second relaxation period is given. This technique is repeated for three times. Three alternate sessions per week is given for 4 weeks.
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Bowen's Technique — In Bowen's Technique, sequence of short gentle moves are applied over Hamstrings. Skin slack is taken to the lateral side of muscle. The muscle is hooked by the thumbs from its lateral edge. Skin is carried along and thumb is flattened in a medial direction, the muscle plucks under the thumbs. Three alternate sessions per week are given for 4 weeks. The treatment time for each session is 20 minutes.
  Arms: Bowen's Technique
Other: Muscle Energy Technique — Isometric contraction of hamstrings is performed by the patient being employing 20% of the strength. This contraction is resisted by the practitioner for 7-10 s. A three second relaxation period is given. This technique is repeated for three times. Three alternate sessions per week is given for 4 weeks.
  Arms: Muscle Energy Technique

SUMMARY:
The aim of this research is to find and compare the effect of Bowen's technique and Muscle energy technique on intensity of pain, active knee extension, limited forward bending and active straight leg raise on hamstrings tightness in patients with chronic non-specific low back pain. A randomized control trial is conducting at Railway General Hospital, Rawalpindi and Al-Ain Hospital, Wah Cantt. The sample size is calculated through open epi is 24. The subjects are divided in two groups, 12 subjects in Bowen's technique group and 12 in Muscle energy technique group. Study duration is of 6 months. Sampling technique applied is non-probability convenient sampling for recruitment and group randomization using sealed envelope method. Only 18-35 years individuals of hamstrings tightness with chronic non-specific low back pain are included. Tools used in the study are Numeric pain rating scale (NPRS), Active knee extension, Sit and reach test, Active straight leg raise and Goniometer. Data will be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Hamstring muscles are well known for their immense tendency to tightness which is due to their multi-joint function, their tonic postural character, and considerable amount of tensional forces to which they are constantly submitted. The ability of the muscle to lengthen allowing one joint (or more than one joint) to move through the range of motion is due to the flexibility of the muscle. If a muscle has good flexibility it will allow muscle tissue to accommodate to imposed stress more easily and allows efficient and effective movement and will assist in preventing or minimizing injuries and enhance performance of the muscle.

The length of the hamstring muscles is considered to play an essential role in both the effectiveness and efficiency of fundamental human movements such as walking and running. Particularly in the field of rehabilitation, flexibility of the muscle is important in postural balance, complete maintenance of the range of motion of knees and hips, injury prevention and optimization of musculoskeletal function. Tight hamstrings have been involved in lumbar spine dysfunction and shows strong positive correlation between low back pain and reduced hamstring flexibility. Hamstring muscle tightness leads to decreased range of motion of lumber flexion and pelvic tilt. This can alter the biomechanics of lumbar spine and may lead to back pain. Mainly hamstrings flexibility may prevent acute and chronic musculoskeletal injuries, low backache problems, postural deviations, gait limitations and chances of fall.

Low back pain (LBP) is described as the pain located in the lower part of the spine (lumbo-sacral region), coming from this area and optionally radiating to one or both lower limbs. It occurs in a great amount of the population, in about 80% of people and it has a different intensity. Non-specific LBP (low back pain) is defined as low back pain not attributable to a known cause there is no pathology within the spine such as cancer, osteoporosis, trauma or fracture. It represents 90-95% of the cases of Low back pain. There are several factors which are responsible for development of Low back pain. Various factors include increased lumber lordosis, reduced abdominal muscle strength, and decreased back extensor muscle endurance, back extensor muscle flexibility, length of iliopsoas and hamstring muscle flexibility.

Muscle energy technique (MET) is a manual technique developed by osteopaths that is now used in much different manual therapy professions. It is gentle manual therapy technique for restricted motion of the spine and extremities and is an active technique where the patient, not the clinician, controls the corrective force.

One of the two techniques is 'Post-isometric relaxation technique (PIRT)' which uses controlled, voluntary isometric contractions up to 20% of a target muscle group. MET is claimed to be useful for lengthening a shortened muscle, improving range of motion at a joint and increasing drainage of fluid from peripheral regions. This approach which targets primarily the soft tissue is also known as 'active muscular relaxation'.

Bowen's technique (BT) was developed by Thomas Bowen in the 1950s in Geelong, Australia which is a dynamic system of muscle and connective tissue therapy. Bowen's Technique is a technique, based on a delicate movement and a series of manipulation of soft tissues. It is a soft tissue therapy, in which therapist uses fingers or thumb to apply gentle rolling moves over muscles, tendons, and other connective tissues in specific parts of the body. Minimum of 2 minutes will be allowed between moves to allow the body to respond and then the whole procedure will be repeated again. Sequence of receiving bilateral moves are applied over segments of erector spinae ,latissimus dorsi, gluteals,the hamstrings muscles proximally and distally, Tenser fascia latae, hip adductors are many more. A classic Bowen's technique session usually lasts from 15 to 45 minutes.

In general, the mechanism of action of Bowen's Technique is based mainly on the concept of proprioception. The skin is innervated tissue and has various types of receptors that detect changes during the position of touch, pressure, vibration, temperature or pain. The fascia also plays the role of a system for collecting, transmitting and processing information. There is even less data on the physiological effects of Bowen's Therapy. There are largely unsubstantiated claims that it acts through effects on fascia, muscle, and cutaneous sensory receptors that give rise to a rebalancing of autonomic nervous system (ANS) activity, muscle relaxation, altered myofibroblast activity, and changes in the type of collagen. Adipocytes and fibroblasts, on the other hand, are responsible for mechano-transduction and lead to a wide range of sensory sensations and communication signals. Therefore, it has been suggested that the contact of the therapist's hands with the patient's skin initiates communication with structures lying deeper. Bowen's studies provide implications of fascially induced following stimulation of mechanoreceptors. The effect of rolling moves that are characteristic of this method is muscular and fascial loosening.

There have been many studies done to check the effectiveness of stretching techniques to increase the flexibility of Hamstrings amongst the most common is MET. Bowen's technique is a specific form of therapy and the concept of treatment of patient according to Bowen's is significantly different from the commonly known methods. There are no studies done pertaining to the comparison of MET and Bowen's Technique for hamstrings flexibility in patients with non-specific low back pain and hence the need of the study arises to check for the more superior form of technique in the treatment of hamstrings flexibility. Until now, the effects of Bowen's Technique therapy have been most often described in the form of a case study. It is difficult to find research conclusions from such works only.

A research was conducted in 2020 entitled as "The effect of muscle energy technique on flexibility of hamstring muscle in Futsal Players" and concluded that Muscle energy technique increased flexibility of hamstrings among futsal players by improving ranges of knee extension. This study also shows the implacability of Muscle Energy Technique in a clinical setting, where it can be performed as a treatment technique for patients who come in for physiotherapy relating to reduced hamstring flexibility.

A research was conducted in 2018 entitled as "Bowen Technique for patients with low back pain" concluded that there were clearly noticeable results in the severity of pain, the range of motion and the degree of disability of respondents referring Oswestry standardized scale. It can be concluded that subsequent treatments would still eliminate pain and improve the health of patients as well.

A research was conducted in 2017 entitled as "Effect of Bowen Technique versus Muscle Energy Technique on Asymptomatic Subjects with Hamstring Tightness" concluded that 3 sessions on alternate days for a week proved to be effective in improving popliteal angle and sit and reach test for flexibility measurements in both Bowen technique as well as muscle energy technique but Bowen technique has shown more improvement in hamstring flexibility and ROM than muscle energy technique.

A research was conducted in 2013 entitled as "Comparative study between the effectiveness of Bowen technique and dynamic soft tissue mobilization in increasing hamstrings flexibility" concluded that there was a significant improvement following the application of Bowen Technique than compared to Dynamic Soft Tissue Mobilization in improving flexibility of hamstring muscle as determined by Active Extension Test.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 degrees active knee extension loss with hip in 90 degree flexion.
* Low back pain from more than 3 months.
* Minimum of 30° restriction in straight leg raise (SLR).
* Currently seeking treatment for low back pain.
* Low back pain radiating above knee.
* Subjects willing to participate in the study.

Exclusion Criteria:

* Fractures of hip and knee.
* SLR greater than 100 degrees.
* Nerve lesion of lower limb.
* Taking medications which may interfere with the results of this study including muscle relaxants.
* Major surgery scheduled during treatment or follow-up period.
* Suspected or conﬁrmed spinal pathology (e.g., tumor, infection, fracture, inﬂammatory disease).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Popliteal angle measurement (active knee extension test) | 12th Day
  Changes from base line ROM range of motion of popliteal angle or active knee extension are taken with the help of goniometer.
NPRS (Numeric Pain rating scale ) | 12th Day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain.
Active Straight Leg Raise (SLR) | 12th Day
  Changes from the Baseline ROM range of Motion of Hip flexion are taken with the Help of Goniometer.
Sit And Reach Test | 12th Day
  Changes from the Baseline measurement are taken with the help of measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srithren NS, Sundaram SS. The Effect of Muscle Energy Technique on Flexibility of Hamstring Muscle in Futsal Players. Malaysian Journal of Movement, Health & Exercise. 2020;9(2).
- [Background] Sailor S, Mehta Y, Shah N, Trivedi A. A comparative study of muscle energy technique and positional release technique on hamstring flexibility in healthy individuals. Journal of Integrated Health Sciences. 2018;6(2):64.
- [Background] Joshi DG, Balthillaya G, Prabhu A. Effect of remote myofascial release on hamstring flexibility in asymptomatic individuals - A randomized clinical trial. J Bodyw Mov Ther. 2018 Jul;22(3):832-837. doi: 10.1016/j.jbmt.2018.01.008. Epub 2018 Feb 17. PMID 30100320
- [Background] Kage V, Bootwala F, Kudchadkar G. Effect of Bowen Technique versus Muscle Energy Technique on Asymptomatic Subjects with Hamstring Tightness: A Randomized Clinical Trial. International Journal of Medical Research & Health Sciences. 2017;6(4):102-8.
- [Background] Lee K, Lewis GN. Short term relief of multisite chronicpain with Bowen Therapy: A double-blind, randomized controlled trial. J Bodyw Mov Ther. 2020 Oct;24(4):271-279. doi: 10.1016/j.jbmt.2020.06.025. Epub 2020 Jul 30. PMID 33218522
- [Background] Banerjee SB, Mukhi S. Immediate Effect of Non Ballistic Active Knee Extension in Neural Slump Position Versus Muscle Energy Technique on Hamstring Flexiblity in Young Adults-Comparitive Study. Indian Journal of Physiotherapy & Occupational Therapy. 2020;14(3):245-52.
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Felix GJS, Black L, Rodrigues M, Silva AG. The acute effect of Bowen therapy on pressure pain thresholds and postural sway in healthy subjects. J Bodyw Mov Ther. 2017 Oct;21(4):804-809. doi: 10.1016/j.jbmt.2016.12.008. Epub 2016 Dec 22. PMID 29037631
- [Background] Ibrahim AA, Akindele MO, Bello B, Kaka B. Translation, Cross-cultural Adaptation, and Psychometric Properties of the Hausa Versions of the Numerical Pain Rating Scale and Global Rating of Change Scale in a Low-literate Population With Chronic Low Back Pain. Spine (Phila Pa 1976). 2020 Apr 15;45(8):E439-E447. doi: 10.1097/BRS.0000000000003306. PMID 31658233
- [Background] Neto T, Jacobsohn L, Carita AI, Oliveira R. Reliability of the Active-Knee-Extension and Straight-Leg-Raise Tests in Subjects With Flexibility Deficits. J Sport Rehabil. 2015 Dec 3;24(4):2014-0220. doi: 10.1123/jsr.2014-0220. Print 2015 Nov 1. PMID 25364856